CLINICAL TRIAL: NCT02151318
Title: Culturing TM Cells From Primary Open-angle Glaucoma Patient Biopsies
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 15309
Record Dates: First submitted 2014-05-21; First posted 2014-05-30 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — The ophthalmologist will collect samples from the tissue that is removed during patients eye surgery that would otherwise be discarded or thrown away. Researchers will collect the sample and grow in the laboratory conditions. These cells will then be studied for further research on glaucoma.
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study, the investigators will collect tissue from patients undergoing trabeculectomy for primary open-angle glaucoma treatment. This tissue would normally be discarded. These trabecular meshwork (TM) cells can be cultured and used experimentally to better understand the mechanisms of glaucoma. These TM biopsies will be cultured on the same day as the trabeculectomy using established techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients having glaucoma and undergoing a trabeculotomy
* Sign ICF (Informed Consent Form)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having glaucoma and undergoing a trabeculotomy
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of new glaucoma medications to reduce TM cellular pathologies associated with the disease glaucoma. | 6 weeks
  TM cell biopsy samples from patients with glaucoma will be harvested and cultured in a laboratory setting to grow primary human TM cells. These cells will be used to test different medications, looking at the medications ability to reduce cellular pathologies commonly seen in TM tissue of patients with glaucoma. Pathologies include myocilin aggregation, and cell death. This will help researchers to determine the most effective compounds in treating glaucoma.

SECONDARY OUTCOMES:
Cultured TM cell toxicity caused by new glaucoma medications | 6 weeks
  Cultured primary TM cells treated with various new medications synthesized to treat cellular pathologies associated with glaucoma, will also be analyzed to look at toxicity caused by the treatments themselves. THis will help to determine the safety of these new medications prior to being administered to patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chad A Dickey, PhD, Principal Investigator — University of South Florida department of Molecular Medicine and Byrd Alzheimer's Institute; Carla Bourne, MD, Study Director — University of South Florida and Tampa General Hospital
Locations (2):
- United States (2):
  - Tampa General Hosipital, Tampa, Florida
  - Byrd Alzheimer's Institute, Tampa, Florida